CLINICAL TRIAL: NCT00005104
Title: Randomized Study of Decreased Hyperinsulinemia on the Ovulatory Response to Clomiphene Citrate in Women With Polycystic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Virginia (Other)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/14915; UVA-HIC-7538; UVA-WSE026
Record Dates: First submitted 2000-04-06; First posted 2000-04-07 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Polycystic Ovary Syndrome; Hyperinsulinism
Keywords: endocrine disorders; hyperinsulinism; polycystic ovarian syndrome; rare disease
MeSH Terms: conditions — Polycystic Ovary Syndrome; Hyperinsulinism; Endocrine System Diseases; Rare Diseases | interventions — Clomiphene; Metformin

INTERVENTIONS:
Drug: clomiphene citrate
Drug: metformin

SUMMARY:
OBJECTIVES:

I. Determine whether reduction of serum insulin levels by metformin increases ovulatory response to clomiphene citrate in women with polycystic ovary syndrome.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double blind, placebo controlled, multicenter study. Patients are randomized to one of two treatment arms.

Patients receive oral metformin or oral placebo three times daily for 7 weeks. Patients remaining anovulatory by day 49 receive metformin or placebo plus escalating doses of oral clomiphene citrate daily for 5 consecutive days, beginning on days 50, 80, and 110. Following ovulation, treatment with clomiphene citrate and metformin or placebo continues until 6 ovulatory cycles occur, pregnancy occurs, or anovulation persists. Patients receiving the placebo arm who have not ovulated on the highest dose of clomiphene citrate may be crossed over to receive metformin after a 6 week washout.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Patients with chronic anovulation due to polycystic ovary syndrome (PCOS) who have failed clomiphene citrate

Must have oligoovulation and hyperandrogenemia

--Prior/Concurrent Therapy--

Endocrine therapy: At least 2 months since prior clomiphene citrate

Other:

* At least 2 months since prior standard therapy (including over the counter drugs)
* At least 2 months since prior investigational drugs
* Prior multi/prenatal vitamins allowed

--Patient Characteristics--

Hematopoietic: Hematocrit greater than 38%

Hepatic:

* Liver function normal
* No clinically significant hepatic disease

Renal:

* No clinically significant renal disease
* Creatinine less than 1.4 mg/dL
* No proteinuria

Cardiovascular: No clinically significant cardiac disease

Pulmonary: No clinically significant pulmonary disease

Hormonal:

* Thyroid function normal
* Prolactin normal
* Estradiol normal
* Fasting 17 alpha-hydroxy progesterone less than 200 ng/dL OR No late onset adrenal hyperplasia 21 alpha-hydroxylase deficiency

Other:

* Not pregnant
* Negative pregnancy test
* Male partner must have a normal semen analysis by WHO criteria
* Must be in acceptable health by interview, medical history, physical exam, and laboratory tests
* No diabetes mellitus
* No clinically significant neurologic, psychiatric, infectious, neoplastic, or metabolic disease
* No clinically significant malignant disease except nonmelanomatous skin cancer
* At least 1 year since any prior drug abuse or alcoholism

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 99
Dates: Start 2000-01

CONTACTS AND LOCATIONS:
Overall Officials: William S. Evans, Study Chair — University of Virginia
Locations (6):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Louisiana State University School of Medicine, Shreveport, Louisiana
  - Washington University - St. Louis, St Louis, Missouri
  - University of Virginia, Charlottesville, Virginia
  - Medical College of Virginia School of Medicine, Richmond, Virginia
- University Alma Mater, Bologna, Italy